CLINICAL TRIAL: NCT03624660
Title: A Phase II Study of Dose-Escalated Proton-Based Radiation Therapy Delivered With a Simultaneous Integrated Boost (SIB) to Intraprostatic Tumors (IPT) Visible on Pretreatment Magnetic Resonance Image
Brief Title: Dose-Escalated Proton Radiation Therapy for High-Risk Prostate Cancer
Acronym: PR11
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB201800933; UFPTI 1712-PR11 (Other: Proton Therapy Institute ID); OCR17697 (Other: Universiy of Florida)
Record Dates: First submitted 2018-07-23; First posted 2018-08-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-05

CONDITIONS: Adenocarcinoma of the Prostate
Keywords: High-risk; Prostate cancer; Proton Radiation; Dose-escalated; Hypofractionation; Simultaneous Integrated Boost (SIB); Intraprostatic Tumor (IPT); Proton Therapy (PT); Androgen Deprivation Therapy (ADT); Magnetic Resonance Imaging (MRI)
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Proton Therapy

STUDY DESIGN:
Intervention Model Description: Patients will be assigned to treatment group according to their lymph node risk or seminal vesicle invasion.
  2 treatment groups:
  * HR-A: Patients with <15% risk of positive pelvic nodes, without posterior extracapsular extension and negative for seminal vesicle invasion on exam pretreatment diagnostic MRI.
  * HR-B: Patient with ≥ 15% risk of positive pelvic nodes or with seminal vesicle invasion, without posterior extracapsular extension.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HR-A (High-risk A) (Experimental): * Prostate and proximal seminal vesicles: 2 cobalt gray equivalent per fraction to a total dose of 78 cobalt gray equivalent.
  * Simultaneous integrated boost to the IPT: 2.2 cobalt gray equivalent per fraction to a total dose of 85.8 cobalt gray equivalent.
  Interventions: Radiation: HR-A
- HR-B (High-risk B) (Experimental): * Prostate, proximal seminal vesicles, and pelvic nodes: 2 cobalt gray equivalent per fraction to a total does of 46 cobalt gray equivalent.
  * Prostate and proximal seminal vesicles: 2 cobalt gray equivalent per fraction to a total dose of 32 cobalt gray equivalent.
  * Entire uninvolved seminal vesicle when part of the seminal vesicle is involved with tumor: 2 cobalt gray equivalent per fraction to a total dose of 78 cobalt gray equivalent.
  * Simultaneous integrated boost to the IPT: 2.2 cobalt gray equivalent per fraction to a total dose of 85.8 cobalt gray equivalent.
  Interventions: Radiation: HR-B

INTERVENTIONS:
Radiation: HR-A — The prostate and proximal seminal vesicles will be treated to 2 cobalt gray equivalent per fraction for 39 fractions for a total of 78 cobalt gray equivalent.
  Simultaneous integrated boost to the IPT will be delivered to 2.2 cobalt gray equivalent per fraction for 39 fractions for a total of 85.8 cobalt gray equivalent.
  Treatment will be given once a day, approximately 5 treatments per week (Monday- Friday), over 8-9 weeks.
  Other Names: Proton Radiation
  Arms: HR-A (High-risk A)
Radiation: HR-B — The prostate, proximal seminal vesicles, and pelvic nodes will be treated to 2 cobalt gray equivalent per fraction for 23 fractions for a total of 46 cobalt gray equivalent.
  The prostate and proximal seminal vesicles will be treated to an additional 2 cobalt gray equivalent per fraction for 16 fractions for a total of 32 cobalt gray equivalent.
  Electively treat the entire uninvolved seminal vesicle to 2 cobalt gray equivalent per fraction for 39 fractions for a total of 78 cobalt gray equivalent when part of the seminal vesicle is involved with tumor.
  Simultaneous integrated boost to the IPT will be delivered to 2.2 cobalt gray equivalent per fraction for 39 fractions for a total of 85.8 cobalt gray equivalent.
  Treatment will be given once a day, approximately 5 treatments per week (Monday- Friday), over 8-9 weeks.
  Other Names: Proton Radiation
  Arms: HR-B (High-risk B)

SUMMARY:
The purpose of this research study is to determine if dose-escalated proton radiation therapy is a good way to treat high-risk prostate cancer. The study features hypofractionation and a simultaneous integrated boost to the magnetic resonance imaging (MRI) identified intraprostatic tumor (IPT) as a method of dose-escalating radiation therapy. The study will include patients with high-risk prostate cancer who are at the highest risk for recurrence. Radiation therapy will be delivered over the course of 8-9 weeks. Additionally, androgen deprivation therapy (ADT) will be started 8-10 weeks prior to starting radiation and continued for a total of 18 months if the patient decides to receive ADT.

DETAILED DESCRIPTION:
Prostate cancer is the most common noncutaneous cancer among men in the United States. The purpose of this research study is to determine if dose-escalated proton radiation therapy is a good way to treat high-risk prostate cancer.

Proton therapy (PT) is a type of ionizing radiation therapy that reduces the dose of excess radiation delivered to normal tissues. By escalating the radiation dose just to the area of the known tumor within the prostate, one could potentially reduce the amount of excess radiation delivered to surrounding organs.This reduction in dose would improve the therapeutic ratio by improving disease control while minimizing the risk for additional toxicity.

In an effort to take advantage of dose escalation's potential for improving disease control but also to limit toxicity, the use of advanced imaging to identify prostate cancer and provide a focal radiation boost to the area have proven to be useful. Recent advances in MRI have made it the most promising technique in identifying and targeting IPTs, improving both cancer control rates and decreasing toxicity.

The study features hypofractionation and a simultaneous integrated boost to the MRI identified intraprostatic tumor (IPT) as a method of dose-escalating radiation therapy. The study will include patients with high-risk prostate cancer who are at the highest risk for recurrence. Radiation therapy will be delivered over the course of 8-9 weeks. Additionally, androgen deprivation therapy (ADT) will be started 8-10 weeks prior to starting radiation and continued for a total of 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient must give study-specific informed consent on an IRB-approved consent prior to any research related procedures or study treatment.
* Patient must be at least 18 years at the time of consent.
* Adenocarcinoma of the prostate with AJCC Clinical Stage T1to T3b disease with histological evaluation via biopsy or repeat biopsy within 12 months prior to registration.
* Patients must undergo a pretreatment diagnostic MRI of the prostate on a 1.5T to 3T Tesla machine within 6 months prior to study registration.
* A focal IPT must be visible on MRI within the prostate and/or seminal vesicles and this MRI must be obtained within 6 months of planning CT scan.
* A biopsy of the dominant lesion is recommended but not required. If an ultrasound guided sextant biopsy was positive for prostatic adenocarcinoma in the area of the MRI identified intraprostatic lesion, this will be acceptable and another guided biopsy targeting the MRI identified disease will not be necessary.
* Patients with at least one of the following high-risk factors: cT3a-T3b OR Gleason 9-10 OR PSA > 30 OR more than 1 high-risk factors must be present: clinical stage of T3, Gleason score 8-10, or PSA 20 ng/ml or greater.
* Hemoglobin must be ≥ 10 g/ml within 4 months prior to registration.
* Zubrod performance status must be 0-1 within 4 months prior to registration.
* If patient has child-producing potential, they must be willing to use medically acceptable contraception during treatment and must be advised to use it for at least 1 year thereafter. This is not applicable if the patient is not sexually active or has had a vasectomy.
* Patients must be able to start treatment within 16 weeks of registration.

Exclusion Criteria:

* T4 prostate disease on CT, MRI, or physical exam.
* Patients unable to undergo MRI of the prostate.
* Patients with a greater than 25% change in prostate volume from the pretreatment MRI of the prostate demonstrating the IPT and the treatment planning MRI. Patients in this case must undergo a repeat diagnostic MRI on a 1.5T to 3.0T Tesla machine and an IPT must still be visible.
* IPT that is more than 75% of the prostate volume when measured on the CT simulation scan.
* Evidence of distant metastasis (M1).
* Patients with positive nodes on cross-sectional imaging.
* Previous prostate cancer local treatment including prostatectomy, hyperthermia, high intensity focused ultrasound, brachytherapy, external-beam radiation therapy, and/or cryotherapy.
* Prior pelvic radiation therapy.
* No prior myocardial infarction within the last 6 months, severe congestive heart failure, or end stage renal disease.
* Active inflammatory bowel disease (diverticulitis, Crohn's disease, ulcerative colitis) affecting the rectum.
* Bilateral hip replacement
* Prior intrapelvic surgery. This includes the following:

  • Bladder surgery
* Prior transurethral resection of the prostate (TURP) or laser ablation for benign prostatic hyperplasia (BPH).
* Patients receiving continuous and current anticoagulation with warfarin sodium (Coumadin), heparin sodium, clopidogrel bisulfate (Plavix), dabigatran etexilate mesylate (Pradaxa), rivaroxaban (Xarelto), apixaban (Eliquis), edoxaban (Savaysa), enoxaparin sodium (Lovenox), prasugrel (Effient), ticagrelor (Brilinta), aspirin/er dipyridamole (Aggrenox), or fondaparinux sodium (Arixtra).

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate cancer is gender-specific. Biological males only.
Enrollment: 100 (Estimated)
Dates: Start 2018-09-24 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Cumulative rate of biochemical failure at 5 years after the end of treatment. | 5 years after the end of radiation therapy
  Biochemical failure will be defined based on the Phoenix definition. Biochemical failure has occurred if the post-treatment prostate-specific antigen (PSA) on at least two occasions rose more than 2 ng/ml above the PSA nadir. Rate of biochemical failure will be measured at 5 years after the end of treatment.

SECONDARY OUTCOMES:
Cumulative rate of acute toxicity observed between day 1 of treatment and 90 days after treatment. | 90 days after the end of radiation therapy
  Assess physician-graded, severe (Grade 3-4), acute (early, within 90 days of treatment) genitourinary and gastrointestinal toxicity rates based on the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Cumulative rate of late toxicity observed between 90 days and 5 years after end of treatment. | 60 months after the end of radiation therapy
  Assess physician-graded, severe (Grade 3-4), late (beginning 90 or more days after treatment), cumulative 5 year genitourinary and gastrointestinal toxicity rates based on the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Rate of change in sexual, bowel, and urinary function from baseline measurement to 5 years after end of treatment. | Rate of change between baseline measurement and 5 years end of radiation therapy
  Assess changes in patient-reported quality of life before and after treatment according to The International Index of Erectile Function (IIEF-5/IIEF-5m) which measures sexual function and the effect of radiation therapy; The International Prostate Symptom Score (IPSS) which measures urinary function and the effect of radiation therapy; and The Expanded Prostate Cancer Index Composite (EPIC) which measures different areas that may be affected by prostate cancer or its treatment.
Assessment of overall and disease-free survival | 5 years after the end of radiation therapy
  Assess the overall survival, defined as the time from the start of treatment to the date of death of any cause, if data is available, at 5 years. Also, cause-specific survival will be calculated.
Assessment of local persistence or local recurrence | 5 years after the end of radiation therapy
  Assess local persistence or local recurrence of prostate cancer at 5 years. Local persistence is defined as the failure of the original abnormal tumor mass seen on cross sectional imaging and/or found on digital rectal exam to resolve in patients who also had a poor PSA response with a PSA nadir greater than 1 ng/mL. Local recurrence is defined as the development of any new abnormal prostate mass on cross sectional imaging or on digital rectal exam with previous exams or imaging showing no mass in the area prior to radiation therapy or after initial treatment.
Rate of distant metastases five years after end of radiation therapy | 5 years after the end of radiation therapy
  Assess the cumulative rate development of distant metastasis up to 5 years after end of radiation. This will be an aggregate binary, yes/no response based on evidence acquired from sources including CT scan, bone scan, and/or PET/CT scan.

CONTACTS AND LOCATIONS:
Overall Officials: Curtis M Bryant, MD, MPH, Principal Investigator — University of Florida Health Proton Therapy Institute
Locations (1):
- University of Florida Health Proton Therapy Institute, Jacksonville, Florida, United States

REFERENCES:
- [Background] American Joint Committee on Cancer. AJCC Cancer Staging Manual. 8thedition ed. New York, NY: Springer; 2017.
- [Background] Bryant C, Smith TL, Henderson RH, Hoppe BS, Mendenhall WM, Nichols RC, Morris CG, Williams CR, Su Z, Li Z, Lee D, Mendenhall NP. Five-Year Biochemical Results, Toxicity, and Patient-Reported Quality of Life After Delivery of Dose-Escalated Image Guided Proton Therapy for Prostate Cancer. Int J Radiat Oncol Biol Phys. 2016 May 1;95(1):422-434. doi: 10.1016/j.ijrobp.2016.02.038. Epub 2016 Feb 16. PMID 27084658
- [Background] Kuban DA, Tucker SL, Dong L, Starkschall G, Huang EH, Cheung MR, Lee AK, Pollack A. Long-term results of the M. D. Anderson randomized dose-escalation trial for prostate cancer. Int J Radiat Oncol Biol Phys. 2008 Jan 1;70(1):67-74. doi: 10.1016/j.ijrobp.2007.06.054. Epub 2007 Aug 31. PMID 17765406
- [Background] Dearnaley DP, Sydes MR, Graham JD, Aird EG, Bottomley D, Cowan RA, Huddart RA, Jose CC, Matthews JH, Millar J, Moore AR, Morgan RC, Russell JM, Scrase CD, Stephens RJ, Syndikus I, Parmar MK; RT01 collaborators. Escalated-dose versus standard-dose conformal radiotherapy in prostate cancer: first results from the MRC RT01 randomised controlled trial. Lancet Oncol. 2007 Jun;8(6):475-87. doi: 10.1016/S1470-2045(07)70143-2. PMID 17482880
- [Background] Zietman AL, Bae K, Slater JD, Shipley WU, Efstathiou JA, Coen JJ, Bush DA, Lunt M, Spiegel DY, Skowronski R, Jabola BR, Rossi CJ. Randomized trial comparing conventional-dose with high-dose conformal radiation therapy in early-stage adenocarcinoma of the prostate: long-term results from proton radiation oncology group/american college of radiology 95-09. J Clin Oncol. 2010 Mar 1;28(7):1106-11. doi: 10.1200/JCO.2009.25.8475. Epub 2010 Feb 1. PMID 20124169
- [Background] Beckendorf V, Guerif S, Le Prise E, Cosset JM, Lefloch O, Chauvet B, Salem N, Chapet O, Bourdin S, Bachaud JM, Maingon P, Lagrange JL, Malissard L, Simon JM, Pommier P, Hay MH, Dubray B, Luporsi E, Bey P. The GETUG 70 Gy vs. 80 Gy randomized trial for localized prostate cancer: feasibility and acute toxicity. Int J Radiat Oncol Biol Phys. 2004 Nov 15;60(4):1056-65. doi: 10.1016/j.ijrobp.2004.05.033. PMID 15519775
- [Background] Rodda S, Tyldesley S, Morris WJ, Keyes M, Halperin R, Pai H, McKenzie M, Duncan G, Morton G, Hamm J, Murray N. ASCENDE-RT: An Analysis of Treatment-Related Morbidity for a Randomized Trial Comparing a Low-Dose-Rate Brachytherapy Boost with a Dose-Escalated External Beam Boost for High- and Intermediate-Risk Prostate Cancer. Int J Radiat Oncol Biol Phys. 2017 Jun 1;98(2):286-295. doi: 10.1016/j.ijrobp.2017.01.008. Epub 2017 Jan 6. PMID 28433432
- [Background] Ippolito E, Mantini G, Morganti AG, Mazzeo E, Padula GD, Digesu C, Cilla S, Frascino V, Luzi S, Massaccesi M, Macchia G, Deodato F, Mattiucci GC, Piermattei A, Cellini N. Intensity-modulated radiotherapy with simultaneous integrated boost to dominant intraprostatic lesion: preliminary report on toxicity. Am J Clin Oncol. 2012 Apr;35(2):158-62. doi: 10.1097/COC.0b013e318209cd8f. PMID 21336090
- [Background] Fonteyne V, Villeirs G, Speleers B, De Neve W, De Wagter C, Lumen N, De Meerleer G. Intensity-modulated radiotherapy as primary therapy for prostate cancer: report on acute toxicity after dose escalation with simultaneous integrated boost to intraprostatic lesion. Int J Radiat Oncol Biol Phys. 2008 Nov 1;72(3):799-807. doi: 10.1016/j.ijrobp.2008.01.040. Epub 2008 Apr 11. PMID 18407430
- [Background] Cellini N, Morganti AG, Mattiucci GC, Valentini V, Leone M, Luzi S, Manfredi R, Dinapoli N, Digesu' C, Smaniotto D. Analysis of intraprostatic failures in patients treated with hormonal therapy and radiotherapy: implications for conformal therapy planning. Int J Radiat Oncol Biol Phys. 2002 Jul 1;53(3):595-9. doi: 10.1016/s0360-3016(02)02795-5. PMID 12062602
- [Background] Pucar D, Hricak H, Shukla-Dave A, Kuroiwa K, Drobnjak M, Eastham J, Scardino PT, Zelefsky MJ. Clinically significant prostate cancer local recurrence after radiation therapy occurs at the site of primary tumor: magnetic resonance imaging and step-section pathology evidence. Int J Radiat Oncol Biol Phys. 2007 Sep 1;69(1):62-9. doi: 10.1016/j.ijrobp.2007.03.065. PMID 17707266
- [Background] Pokorny MR, de Rooij M, Duncan E, Schroder FH, Parkinson R, Barentsz JO, Thompson LC. Prospective study of diagnostic accuracy comparing prostate cancer detection by transrectal ultrasound-guided biopsy versus magnetic resonance (MR) imaging with subsequent MR-guided biopsy in men without previous prostate biopsies. Eur Urol. 2014 Jul;66(1):22-9. doi: 10.1016/j.eururo.2014.03.002. Epub 2014 Mar 14. PMID 24666839
- [Background] Van Vulpen M, Van Loon J, Pos F, et al. OC-0282: FLAME randomised trial: 95Gy MRI-boost vs 77Gy prostate radiotherapy: toxicity and quality of life. Radiother Oncol. 2016;119(1 Suppl):S132.
- [Background] Pollack A, Walker G, Horwitz EM, Price R, Feigenberg S, Konski AA, Stoyanova R, Movsas B, Greenberg RE, Uzzo RG, Ma C, Buyyounouski MK. Randomized trial of hypofractionated external-beam radiotherapy for prostate cancer. J Clin Oncol. 2013 Nov 1;31(31):3860-8. doi: 10.1200/JCO.2013.51.1972. Epub 2013 Oct 7. PMID 24101042
- [Background] American Cancer Society. Cancer Facts & Figures 2016. 2016; https://www.cancer.org/research/cancer-facts-statistics/all-cancer-facts-figures/cancer-facts-figures-2016.html. Accessed 10/03/2017.
- [Background] Chism DB, Hanlon AL, Horwitz EM, Feigenberg SJ, Pollack A. A comparison of the single and double factor high-risk models for risk assignment of prostate cancer treated with 3D conformal radiotherapy. Int J Radiat Oncol Biol Phys. 2004 Jun 1;59(2):380-5. doi: 10.1016/j.ijrobp.2003.10.059. PMID 15145151
- [Background] Roach M, Lu J, Pilepich MV, Asbell SO, Mohiuddin M, Terry R, Grignon D. Four prognostic groups predict long-term survival from prostate cancer following radiotherapy alone on Radiation Therapy Oncology Group clinical trials. Int J Radiat Oncol Biol Phys. 2000 Jun 1;47(3):609-15. doi: 10.1016/s0360-3016(00)00578-2. PMID 10837943
- [Background] D'Amico AV, Whittington R, Malkowicz SB, Cote K, Loffredo M, Schultz D, Chen MH, Tomaszewski JE, Renshaw AA, Wein A, Richie JP. Biochemical outcome after radical prostatectomy or external beam radiation therapy for patients with clinically localized prostate carcinoma in the prostate specific antigen era. Cancer. 2002 Jul 15;95(2):281-6. doi: 10.1002/cncr.10657. PMID 12124827
- [Background] National Comprehensive Cancer Network. NCCN Clinical Practice Guidelines in Oncology: Prostate Cancer. 2017; https://www.nccn.org/professionals/physician_gls/PDF/prostate.pdf. Accessed 10/03/2017.
- [Background] Nguyen QN, Levy LB, Lee AK, Choi SS, Frank SJ, Pugh TJ, McGuire S, Hoffman K, Kuban DA. Long-term outcomes for men with high-risk prostate cancer treated definitively with external beam radiotherapy with or without androgen deprivation. Cancer. 2013 Sep 15;119(18):3265-71. doi: 10.1002/cncr.28213. Epub 2013 Jun 24. PMID 23798338
- [Background] Spratt DE, Pei X, Yamada J, Kollmeier MA, Cox B, Zelefsky MJ. Long-term survival and toxicity in patients treated with high-dose intensity modulated radiation therapy for localized prostate cancer. Int J Radiat Oncol Biol Phys. 2013 Mar 1;85(3):686-92. doi: 10.1016/j.ijrobp.2012.05.023. Epub 2012 Jul 12. PMID 22795805
- [Background] Aizer AA, Yu JB, Colberg JW, McKeon AM, Decker RH, Peschel RE. Radical prostatectomy vs. intensity-modulated radiation therapy in the management of localized prostate adenocarcinoma. Radiother Oncol. 2009 Nov;93(2):185-91. doi: 10.1016/j.radonc.2009.09.001. Epub 2009 Oct 1. PMID 19800702
- [Background] Vora SA, Wong WW, Schild SE, Ezzell GA, Andrews PE, Ferrigni RG, Swanson SK. Outcome and toxicity for patients treated with intensity modulated radiation therapy for localized prostate cancer. J Urol. 2013 Aug;190(2):521-6. doi: 10.1016/j.juro.2013.02.012. Epub 2013 Feb 13. PMID 23415964
- [Background] Morris WJ, Tyldesley S, Rodda S, Halperin R, Pai H, McKenzie M, Duncan G, Morton G, Hamm J, Murray N. Androgen Suppression Combined with Elective Nodal and Dose Escalated Radiation Therapy (the ASCENDE-RT Trial): An Analysis of Survival Endpoints for a Randomized Trial Comparing a Low-Dose-Rate Brachytherapy Boost to a Dose-Escalated External Beam Boost for High- and Intermediate-risk Prostate Cancer. Int J Radiat Oncol Biol Phys. 2017 Jun 1;98(2):275-285. doi: 10.1016/j.ijrobp.2016.11.026. Epub 2016 Nov 24. PMID 28262473
- [Background] Haustermans KM, Hofland I, Van Poppel H, Oyen R, Van de Voorde W, Begg AC, Fowler JF. Cell kinetic measurements in prostate cancer. Int J Radiat Oncol Biol Phys. 1997 Mar 15;37(5):1067-70. doi: 10.1016/s0360-3016(96)00579-2. PMID 9169814
- [Background] Duchesne GM, Peters LJ. What is the alpha/beta ratio for prostate cancer? Rationale for hypofractionated high-dose-rate brachytherapy. Int J Radiat Oncol Biol Phys. 1999 Jul 1;44(4):747-8. doi: 10.1016/s0360-3016(99)00024-3. No abstract available. PMID 10386630
- [Background] Dasu A, Toma-Dasu I. Prostate alpha/beta revisited -- an analysis of clinical results from 14 168 patients. Acta Oncol. 2012 Nov;51(8):963-74. doi: 10.3109/0284186X.2012.719635. Epub 2012 Sep 12. PMID 22966812
- [Background] Miralbell R, Roberts SA, Zubizarreta E, Hendry JH. Dose-fractionation sensitivity of prostate cancer deduced from radiotherapy outcomes of 5,969 patients in seven international institutional datasets: alpha/beta = 1.4 (0.9-2.2) Gy. Int J Radiat Oncol Biol Phys. 2012 Jan 1;82(1):e17-24. doi: 10.1016/j.ijrobp.2010.10.075. Epub 2011 Feb 15. PMID 21324610
- [Background] Brenner DJ, Hall EJ. Fractionation and protraction for radiotherapy of prostate carcinoma. Int J Radiat Oncol Biol Phys. 1999 Mar 15;43(5):1095-101. doi: 10.1016/s0360-3016(98)00438-6. PMID 10192361
- [Background] Brenner DJ. Fractionation and late rectal toxicity. Int J Radiat Oncol Biol Phys. 2004 Nov 15;60(4):1013-5. doi: 10.1016/j.ijrobp.2004.04.014. No abstract available. PMID 15519768
- [Background] Tucker SL, Thames HD, Michalski JM, Bosch WR, Mohan R, Winter K, Cox JD, Purdy JA, Dong L. Estimation of alpha/beta for late rectal toxicity based on RTOG 94-06. Int J Radiat Oncol Biol Phys. 2011 Oct 1;81(2):600-5. doi: 10.1016/j.ijrobp.2010.11.080. Epub 2011 Mar 4. PMID 21377288
- [Background] Michalski JM, Moughan J, Purdy JA, et al. Initial Results of a Phase 3 Randomized Study of High Dose 3DCRT/IMRT versus Standard Dose 3D-CRT/IMRT in Patients Treated for Localized Prostate Cancer (RTOG 0126). Int J Radiat Oncol Biol Phys. 2014;90(5):1263.
- [Background] Beckendorf V, Guerif S, Le Prise E, Cosset JM, Bougnoux A, Chauvet B, Salem N, Chapet O, Bourdain S, Bachaud JM, Maingon P, Hannoun-Levi JM, Malissard L, Simon JM, Pommier P, Hay M, Dubray B, Lagrange JL, Luporsi E, Bey P. 70 Gy versus 80 Gy in localized prostate cancer: 5-year results of GETUG 06 randomized trial. Int J Radiat Oncol Biol Phys. 2011 Jul 15;80(4):1056-63. doi: 10.1016/j.ijrobp.2010.03.049. Epub 2010 Dec 14. PMID 21147514
- [Background] Weinreb JC, Barentsz JO, Choyke PL, Cornud F, Haider MA, Macura KJ, Margolis D, Schnall MD, Shtern F, Tempany CM, Thoeny HC, Verma S. PI-RADS Prostate Imaging - Reporting and Data System: 2015, Version 2. Eur Urol. 2016 Jan;69(1):16-40. doi: 10.1016/j.eururo.2015.08.052. Epub 2015 Oct 1. PMID 26427566
- [Background] Woo S, Suh CH, Kim SY, Cho JY, Kim SH. Diagnostic Performance of Prostate Imaging Reporting and Data System Version 2 for Detection of Prostate Cancer: A Systematic Review and Diagnostic Meta-analysis. Eur Urol. 2017 Aug;72(2):177-188. doi: 10.1016/j.eururo.2017.01.042. Epub 2017 Feb 11. PMID 28196723
- [Background] Vargas C, Fryer A, Mahajan C, Indelicato D, Horne D, Chellini A, McKenzie C, Lawlor P, Henderson R, Li Z, Lin L, Olivier K, Keole S. Dose-volume comparison of proton therapy and intensity-modulated radiotherapy for prostate cancer. Int J Radiat Oncol Biol Phys. 2008 Mar 1;70(3):744-51. doi: 10.1016/j.ijrobp.2007.07.2335. Epub 2007 Sep 27. PMID 17904306
- [Background] Chera BS, Vargas C, Morris CG, Louis D, Flampouri S, Yeung D, Duvvuri S, Li Z, Mendenhall NP. Dosimetric study of pelvic proton radiotherapy for high-risk prostate cancer. Int J Radiat Oncol Biol Phys. 2009 Nov 15;75(4):994-1002. doi: 10.1016/j.ijrobp.2009.01.044. Epub 2009 Jul 18. PMID 19619961
- [Background] Hoppe BS, Michalski JM, Mendenhall NP, Morris CG, Henderson RH, Nichols RC, Mendenhall WM, Williams CR, Regan MM, Chipman JJ, Crociani CM, Sandler HM, Sanda MG, Hamstra DA. Comparative effectiveness study of patient-reported outcomes after proton therapy or intensity-modulated radiotherapy for prostate cancer. Cancer. 2014 Apr 1;120(7):1076-82. doi: 10.1002/cncr.28536. Epub 2013 Dec 30. PMID 24382757
- [Background] Mendenhall NP, Li Z, Hoppe BS, Marcus RB Jr, Mendenhall WM, Nichols RC, Morris CG, Williams CR, Costa J, Henderson R. Early outcomes from three prospective trials of image-guided proton therapy for prostate cancer. Int J Radiat Oncol Biol Phys. 2012 Jan 1;82(1):213-21. doi: 10.1016/j.ijrobp.2010.09.024. Epub 2010 Nov 17. PMID 21093164
- [Background] Slater JD, Rossi CJ Jr, Yonemoto LT, Bush DA, Jabola BR, Levy RP, Grove RI, Preston W, Slater JM. Proton therapy for prostate cancer: the initial Loma Linda University experience. Int J Radiat Oncol Biol Phys. 2004 Jun 1;59(2):348-52. doi: 10.1016/j.ijrobp.2003.10.011. PMID 15145147
- [Background] Liauw SL, Weichselbaum RR, Rash C, Correa D, Al-Hallaq HA, Pelizzari CA, Jani AB. Biochemical control and toxicity after intensity-modulated radiation therapy for prostate cancer. Technol Cancer Res Treat. 2009 Jun;8(3):201-6. doi: 10.1177/153303460900800304. PMID 19445537
- [Background] Pugh TJ, Munsell MF, Choi S, Nguyen QN, Mathai B, Zhu XR, Sahoo N, Gillin M, Johnson JL, Amos RA, Dong L, Mahmood U, Kuban DA, Frank SJ, Hoffman KE, McGuire SE, Lee AK. Quality of life and toxicity from passively scattered and spot-scanning proton beam therapy for localized prostate cancer. Int J Radiat Oncol Biol Phys. 2013 Dec 1;87(5):946-53. doi: 10.1016/j.ijrobp.2013.08.032. Epub 2013 Oct 15. PMID 24139077
- [Background] Briganti A, Larcher A, Abdollah F, Capitanio U, Gallina A, Suardi N, Bianchi M, Sun M, Freschi M, Salonia A, Karakiewicz PI, Rigatti P, Montorsi F. Updated nomogram predicting lymph node invasion in patients with prostate cancer undergoing extended pelvic lymph node dissection: the essential importance of percentage of positive cores. Eur Urol. 2012 Mar;61(3):480-7. doi: 10.1016/j.eururo.2011.10.044. Epub 2011 Nov 7. PMID 22078338
- [Background] Yu JB, Makarov DV, Gross C. A new formula for prostate cancer lymph node risk. Int J Radiat Oncol Biol Phys. 2011 May 1;80(1):69-75. doi: 10.1016/j.ijrobp.2010.01.068. Epub 2010 Jun 30. PMID 20594769
- [Background] Eifler JB, Feng Z, Lin BM, Partin MT, Humphreys EB, Han M, Epstein JI, Walsh PC, Trock BJ, Partin AW. An updated prostate cancer staging nomogram (Partin tables) based on cases from 2006 to 2011. BJU Int. 2013 Jan;111(1):22-9. doi: 10.1111/j.1464-410X.2012.11324.x. Epub 2012 Jul 26. PMID 22834909
- [Background] Lawton CA, DeSilvio M, Roach M 3rd, Uhl V, Kirsch R, Seider M, Rotman M, Jones C, Asbell S, Valicenti R, Hahn S, Thomas CR Jr. An update of the phase III trial comparing whole pelvic to prostate only radiotherapy and neoadjuvant to adjuvant total androgen suppression: updated analysis of RTOG 94-13, with emphasis on unexpected hormone/radiation interactions. Int J Radiat Oncol Biol Phys. 2007 Nov 1;69(3):646-55. doi: 10.1016/j.ijrobp.2007.04.003. Epub 2007 May 24. PMID 17531401
- [Background] Roach M 3rd, Bae K, Speight J, Wolkov HB, Rubin P, Lee RJ, Lawton C, Valicenti R, Grignon D, Pilepich MV. Short-term neoadjuvant androgen deprivation therapy and external-beam radiotherapy for locally advanced prostate cancer: long-term results of RTOG 8610. J Clin Oncol. 2008 Feb 1;26(4):585-91. doi: 10.1200/JCO.2007.13.9881. Epub 2008 Jan 2. PMID 18172188
- [Background] Bolla M, Van Tienhoven G, Warde P, Dubois JB, Mirimanoff RO, Storme G, Bernier J, Kuten A, Sternberg C, Billiet I, Torecilla JL, Pfeffer R, Cutajar CL, Van der Kwast T, Collette L. External irradiation with or without long-term androgen suppression for prostate cancer with high metastatic risk: 10-year results of an EORTC randomised study. Lancet Oncol. 2010 Nov;11(11):1066-73. doi: 10.1016/S1470-2045(10)70223-0. Epub 2010 Oct 7. PMID 20933466
- [Background] Denham JW, Steigler A, Lamb DS, Joseph D, Turner S, Matthews J, Atkinson C, North J, Christie D, Spry NA, Tai KH, Wynne C, D'Este C. Short-term neoadjuvant androgen deprivation and radiotherapy for locally advanced prostate cancer: 10-year data from the TROG 96.01 randomised trial. Lancet Oncol. 2011 May;12(5):451-9. doi: 10.1016/S1470-2045(11)70063-8. PMID 21440505
- [Background] D'Amico AV, Manola J, Loffredo M, Renshaw AA, DellaCroce A, Kantoff PW. 6-month androgen suppression plus radiation therapy vs radiation therapy alone for patients with clinically localized prostate cancer: a randomized controlled trial. JAMA. 2004 Aug 18;292(7):821-7. doi: 10.1001/jama.292.7.821. PMID 15315996
- [Background] Horwitz EM, Bae K, Hanks GE, Porter A, Grignon DJ, Brereton HD, Venkatesan V, Lawton CA, Rosenthal SA, Sandler HM, Shipley WU. Ten-year follow-up of radiation therapy oncology group protocol 92-02: a phase III trial of the duration of elective androgen deprivation in locally advanced prostate cancer. J Clin Oncol. 2008 May 20;26(15):2497-504. doi: 10.1200/JCO.2007.14.9021. Epub 2008 Apr 14. PMID 18413638
- [Background] Nabid A, Carrier N, Martin AG, Bahary JP, Lemaire C, Vass S, Bahoric B, Archambault R, Vincent F, Bettahar R, Duclos M, Garant MP, Souhami L. Duration of Androgen Deprivation Therapy in High-risk Prostate Cancer: A Randomized Phase III Trial. Eur Urol. 2018 Oct;74(4):432-441. doi: 10.1016/j.eururo.2018.06.018. Epub 2018 Jul 3. PMID 29980331
- [Background] Pilepich MV, Winter K, Lawton CA, Krisch RE, Wolkov HB, Movsas B, Hug EB, Asbell SO, Grignon D. Androgen suppression adjuvant to definitive radiotherapy in prostate carcinoma--long-term results of phase III RTOG 85-31. Int J Radiat Oncol Biol Phys. 2005 Apr 1;61(5):1285-90. doi: 10.1016/j.ijrobp.2004.08.047. PMID 15817329
- [Background] Bolla M, de Reijke TM, Van Tienhoven G, Van den Bergh AC, Oddens J, Poortmans PM, Gez E, Kil P, Akdas A, Soete G, Kariakine O, van der Steen-Banasik EM, Musat E, Pierart M, Mauer ME, Collette L; EORTC Radiation Oncology Group and Genito-Urinary Tract Cancer Group. Duration of androgen suppression in the treatment of prostate cancer. N Engl J Med. 2009 Jun 11;360(24):2516-27. doi: 10.1056/NEJMoa0810095. PMID 19516032
- [Background] Ghilezan MJ, Jaffray DA, Siewerdsen JH, Van Herk M, Shetty A, Sharpe MB, Zafar Jafri S, Vicini FA, Matter RC, Brabbins DS, Martinez AA. Prostate gland motion assessed with cine-magnetic resonance imaging (cine-MRI). Int J Radiat Oncol Biol Phys. 2005 Jun 1;62(2):406-17. doi: 10.1016/j.ijrobp.2003.10.017. PMID 15890582
- [Background] Padhani AR, Khoo VS, Suckling J, Husband JE, Leach MO, Dearnaley DP. Evaluating the effect of rectal distension and rectal movement on prostate gland position using cine MRI. Int J Radiat Oncol Biol Phys. 1999 Jun 1;44(3):525-33. doi: 10.1016/s0360-3016(99)00040-1. PMID 10348281
- [Background] Litzenberg DW, Balter JM, Hadley SW, Sandler HM, Willoughby TR, Kupelian PA, Levine L. Influence of intrafraction motion on margins for prostate radiotherapy. Int J Radiat Oncol Biol Phys. 2006 Jun 1;65(2):548-53. doi: 10.1016/j.ijrobp.2005.12.033. Epub 2006 Mar 20. PMID 16545919
- [Background] Litzenberg D, Dawson LA, Sandler H, Sanda MG, McShan DL, Ten Haken RK, Lam KL, Brock KK, Balter JM. Daily prostate targeting using implanted radiopaque markers. Int J Radiat Oncol Biol Phys. 2002 Mar 1;52(3):699-703. doi: 10.1016/s0360-3016(01)02654-2. PMID 11849792
- [Background] Vargas C, Yan D, Kestin LL, Krauss D, Lockman DM, Brabbins DS, Martinez AA. Phase II dose escalation study of image-guided adaptive radiotherapy for prostate cancer: use of dose-volume constraints to achieve rectal isotoxicity. Int J Radiat Oncol Biol Phys. 2005 Sep 1;63(1):141-9. doi: 10.1016/j.ijrobp.2004.12.017. PMID 16111582
- See also: Contact the University of Florida Health Proton Therapy Institute — https://www.floridaproton.org/about-us/contact-us